CLINICAL TRIAL: NCT05089890
Title: An Open, Single-centre, Clinical Investigation to Explore the Binding of Bacteria and Fungi to Dialkylcarbamoyl Chloride (DACC)-Coated Dressings From Hard-to-heal Wounds
Brief Title: Clinical Investigation of Sorbact® Dressings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ABIGO Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DHF-5474
Record Dates: First submitted 2021-09-30; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Hard-to-heal Wounds; Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer; Arterial Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The patients will be divided in 3 cohorts and will be treated with 3 different devices. The choice of which dressing to use depends of the characters of the wounds.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sorbact® Compress (Other): Patients already assigned to start treatment with Sorbact® Compress as it is judged by the investigator to be the most suitable for their wounds
  Interventions: Device: Sorbact® Compress
- Sorbact® Gel Dressing (Other): Patients already assigned to start treatment with Sorbact® Gel Dressing as it is judged by the investigator to be the most suitable for their wounds
  Interventions: Device: Sorbact® Gel Dressing
- Sorbact® Ribbon Gauze (Other): Patients already assigned to start treatment with Sorbact® Ribbon Gauze as it is judged by the investigator to be the most suitable for their wounds
  Interventions: Device: Sorbact® Ribbon Gauze

INTERVENTIONS:
Device: Sorbact® Compress — Sorbact® technology is a bacteria- and fungi-binding wound contact layer from which Sorbact® Compress has been developed. The patients will be in one of these 3 arms depending on the choice of dressing most suitable for their wounds.
  The purpose of the study is not to compare between the devices, but to study each device on its own.
  Arms: Sorbact® Compress
Device: Sorbact® Gel Dressing — Sorbact® technology is a bacteria- and fungi-binding wound contact layer from which Sorbact® Gel Dressing has been developed. The patients will be in one of these 3 arms depending on the choice of dressing most suitable for their wounds.
  The purpose of the study is not to compare between the devices, but to study each device on its own.
  Arms: Sorbact® Gel Dressing
Device: Sorbact® Ribbon Gauze — Sorbact® technology is a bacteria- and fungi-binding wound contact layer from which Sorbact® Ribbon Gauze has been developed. The patients will be in one of these 3 arms depending on the choice of dressing most suitable for their wounds.
  The purpose of the study is not to compare between the devices, but to study each device on its own.
  Arms: Sorbact® Ribbon Gauze

SUMMARY:
The main purpose of this exploratory clinical investigation is to study the binding of bacteria and fungi from hard-to-heal wounds to the DACC-coated dressings.

DETAILED DESCRIPTION:
This is a prospective, open, single-centre, exploratory clinical investigation with a primary objective of studying the binding of bacteria and fungi from hard-to-heal wounds to the surface of DACC-coated dressings.

Subjects suffering from hard-to-heal wounds who are due to start using a dressing from the Sorbact range will be recruited at one investigation site in Sweden. The subjects will be divided into three groups by dressing type and there will be 10 subjects in each group, i.e., 10 subjects will be treated with Sorbact® Compress, 10 subjects will be treated with Sorbact® Gel Dressing, and 10 subjects will be treated with Sorbact® Ribbon Gauze. The dressings will be used in accordance with their respective IFU.

The clinical investigation is designed to have a treatment period of 14 days with no additional follow-up.

Three visits are planned for each subject, including a screening/baseline visit at the clinic and two further visits to the study clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the Subject Information and Informed Consent Form and provide meaningful informed consent
2. Due to start using one of the following dressings: Sorbact® Compress, Sorbact® Gel Dressing and Sorbact® Ribbon Gauze
3. Age ≥18 years
4. Presence of hard-to-heal wound for ≥6 weeks with no significant wound area reduction for the last 4 weeks confirmed by investigator/study nurse

Exclusion Criteria:

1. Participating in another clinical investigation
2. Known allergy or sensitivity to any components of the allocated investigational device
3. Use of systemic or topical antibiotic for the past two weeks or planning to use while participating in investigation.
4. Use of antimicrobial agent (e.g., silver- or iodine-containing dressings, or gels) during the last wo weeks
5. Use of a dressing from the Sorbact® range during the last two weeks
6. Subjects with any other condition that as judged by the investigator may make investigation procedures inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Bacterial and fungal species irreversibly bound to the dressing after 2 days (+ 1 day). | 2 days (+1 day)
  The measurements that will be used to assess the primary outcome are 16S rRNA sequencing to identify bacterial species, Internal Transcribed Spacer (ITS) sequencing to identify fungal species and scanning electron microscopy (SEM) images for visualization of bacteria and fungi bound to the dressing

SECONDARY OUTCOMES:
Wound bed microbial load at 14 days (±1 days) compared to baseline | 14 days (±1 days)
  qPCR (quantitiative polymerase chain reaction) will be used.
Wound bed bacteria and fungi species at baseline and at 14 days (±1 days) | 14 days (±1 days)
  16S rRNA and Internal Transcribed Spacer (ITS) sequencing will be used.
Presence of endotoxin on the dressing after 2 days (+ 1 day) | 2 days (+ 1 day)
  LAL (Limulus amoebocyt lysat) method will be used.
Wound fluid endotoxin level at 14 days (±1 days) compared to baseline | 14 days (±1 days)
  LAL (Limulus amoebocyt lysat) method will be used.
Presence of inflammatory biomarkers on the dressing after 2 days (+ 1 day) | 2 days (+ 1 day)
  PEA (proximity extension assay) will be used.
Wound fluid inflammatory biomarker levels at 14 days (±1 days) compared to baseline | 14 days (±1 days)
  PEA (proximity extension assay) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jönsson, MD, Principal Investigator — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No